CLINICAL TRIAL: NCT02592577
Title: A Phase I Dose Escalation Open Label Clinical Trial Evaluating the Safety and Efficacy of MAGE A10ᶜ⁷⁹⁶T in Subjects With Stage IIIb or Stage IV Non-Small Cell Lung Cancer (NSCLC)
Brief Title: MAGE A10ᶜ⁷⁹⁶T for Advanced NSCLC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adaptimmune (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADP 0022-003
Record Dates: First submitted 2015-10-20; First posted 2015-10-30 (Estimated); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Non-Small Cell Lung Cancer; Carcinoma
Keywords: Previously Treated; Cell Therapy; T Cell Therapy; MAGE-A10; Immuno-oncology; T Cell Receptor; Metastatic
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Autologous Genetically modified T cells, MAGEA10ᶜ⁷⁹⁶T (Experimental)
  Interventions: Biological: Autologous Genetically modified T cells, MAGEA10ᶜ⁷⁹⁶T

INTERVENTIONS:
Biological: Autologous Genetically modified T cells, MAGEA10ᶜ⁷⁹⁶T

SUMMARY:
This first time in human study is intended for men and women at least 18 years of age who have advanced lung cancer which has grown or returned after being treated. In particular, it is a study for subjects who have a blood test positive for HLA-A*02:01 and/or HLA-A*02:06 and a tumor test positive for MAGE A10 protein expression (protein or gene). This trial is a dose escalation trial that will evaluate 3 doses of transduced cells administered after a lymphodepleting chemotherapy regimen using a 3+3 dose escalation design .The study will take the subject's T cells, which are a natural type of immune cell in the blood, and send them to a laboratory to be modified. The changed T cells used in this study will be the subject's own T cells that have been genetically changed with the aim of attacking and destroying cancer cells.

When the MAGE A10ᶜ⁷⁹⁶T cells are available, subjects will receive lymphodepleting chemotherapy with cyclophosphamide and fludarabine, followed by the T cell infusion. The purpose of this study is to test the safety of genetically changed T cells and find out what effects, if any, they have in subjects with lung cancer. The study will evaluate three different cell dose levels in order to find out the target cell dose. Once the target cell dose is determined, additional subjects will be enrolled to further test the safety and effects at this cell dose.

Subjects will be seen frequently by the Study Physician right after receiving their T cells back and up to first 6 months. After that, subjects will be seen every three months. Subjects will be seen every 6 months by their Study Physician for the first 5 years after the T cell infusion. If the T cells are found in the blood at five years, then the subjects will continue to be seen once a year until the T cells are no longer found in the blood for a maximum of 15 years. If the T cells are no longer found in the blood at 5 years, then the subject will be contacted by the Study Physician for the next 10 years. Subjects who have a confirmed response or clinical benefit ≥4 weeks after the first T-cell infusion and whose tumor continues to express the appropriate antigen target may be eligible for a second infusion. All subjects, completing or withdrawing from the Interventional Phase of the study, will enter a 15-year long-term follow-up phase for observation of delayed adverse events. All subjects will continue to be followed for overall survival during the long-term follow-up phase.

ELIGIBILITY:
Key Inclusion Criteria:

1. Subject has histologically or cytologically confirmed diagnosis of advanced non-small cell lung cancer (stage IIIB or IV) or recurrent disease
2. Subject has received at least one line of prior therapy
3. Subjects with known epidermal growth factor receptor (EGFR) mutations or anaplastic lymphoma kinase receptor (ALK) or ROS1 gene rearrangements must have failed (progressive disease or unacceptable toxicity) at least one prior EGFR or ALK or ROS1 tyrosine kinase inhibitor, respectively. Subject may have received PD-1 or PDL-1 inhibitors and or chemotherapy. There is no limit on lines of prior anti-cancer therapy (a washout period applies for recent anti-cancer treatments).
4. Subject has measurable disease according to RECIST v1.1 criteria prior to lymphodepletion.
5. Subject is HLA-A*02:01 or HLA-A*02:06 positive.
6. Subject's tumor (either an archival specimen or a fresh biopsy if archival tissue is unavailable) has been pathologically reviewed by a designated central laboratory confirming MAGE-A10 expression.
7. Subject has an ECOG Performance Status 0-1 and anticipated life expectancy >6 months prior to apheresis and >3 months prior to lymphodepletion.
8. Subject is ≥18 to ≤75 years of age
9. Adequate organ function

Key Exclusion Criteria:

1. Subject is HLA-A*02:05, HLA-B*15:01 and/or HLA-B*46:01 positive.
2. History of chronic or recurrent (within the last year prior to enrollment) severe autoimmune or active immune-mediated disease requiring steroids or other immunosuppressive treatments.
3. Subject has symptomatic CNS metastases. Subjects with prior history of symptomatic CNS metastasis must have received treatment and be neurologically stable for at least 1 month prior to leukapheresis and lymphodepletion.
4. Active malignancy besides NSCLC within 3 years prior to screening.
5. Uncontrolled intercurrent illness including, but not limited to:

   * Ongoing or active infection;
   * Clinically significant cardiac disease
   * Inadequate pulmonary function
   * Interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2021-03-17 (Actual)

PRIMARY OUTCOMES:
Number of subjects with dose-limiting toxicity (DLT) and adverse events (AE), including serious adverse events (SAE) | 24 months
  Determine if treatment with autologous genetically modified T cells, (MAGE A10ᶜ⁷⁹⁶T ) is safe and tolerable through assessment of DLTs, AEs, including SAEs; laboratory assessments, including chemistry, hematology, and coagulation; cardiac and pulmonary assessments, including ECG and troponin.

SECONDARY OUTCOMES:
Proportion of subjects with a confirmed Complete Response (CR) or Partial Response (PR) | 24 months
  Evaluation of the efficacy of the treatment by assessment of the Overall Response Rate according to RECIST v1.1
Interval between the date of first T cell infusion dose and first documented evidence of CR or PR | 24 months
  Evaluation of the efficacy of the treatment by assessment of time to first response
Interval between the date of first documented evidence of CR or PR until first documented disease progression or death due to any cause | 24 months
  Evaluation of the efficacy of the treatment by assessment of duration of response
Interval between the date of first documented evidence of SD until first documented disease progression or death due to any cause | 24 months
  Evaluation of the efficacy of the treatment by assessment of duration of stable disease
Interval between the date of first T cell infusion and the earliest date of disease progression or death due to any cause | 24 months
  Evaluation of the efficacy of the treatment by assessment of progression-free survival
Interval between the date of first T cell infusion and date of disease progression or death due to any cause | 24 months
  Evaluation of the efficacy of the treatment by assessment of overall survival
Best Overall Response (BOR) | 24 months
  Best Overall Response (BOR), defined as the best response recorded from the date of T cell infusion until disease progression
To evaluate potential gene therapy-related delayed adverse events for 15 years post infusion. | 15 years
  Presence of any of the following LTFU AEs:
  * New malignancies
  * New incidence or exacerbation of a pre-existing neurologic disorder
  * New incidence or exacerbation of a prior rheumatologic or other autoimmune disorder
  * New incidence of a hematologic disorder
  * Opportunistic and/or serious infections
  * Unanticipated illness and/or hospitalization deemed related to gene modified cell therapy Persistence of MAGE-A10c796T and replication-competent lentivirus (RCL) over time.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Creelan, MD, MS, Study Chair — H. Lee Moffitt Cancer Center
Locations (19):
- United States (14):
  - City of Hope, Duarte, California
  - Stanford Cancer Center, Palo Alto, California
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - University of Maryland, Greenebaum Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University, School of Medicine, St Louis, Missouri
  - Duke University Medical Center, Duke Cancer Institute, Durham, North Carolina
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Tennessee Oncology- Sarah Cannon Research Institute, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- Spain (2):
  - Hospital Universitario Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Universitario 12 Octubre Avda. de Córdoba s/n, Madrid, Madrid
- United Kingdom (2):
  - University College Hospital Macmillan Cancer Centre, London
  - The Christie NHS Foundation Trust, Manchester

REFERENCES:
- [Derived] Blumenschein GR, Devarakonda S, Johnson M, Moreno V, Gainor J, Edelman MJ, Heymach JV, Govindan R, Bachier C, Doger de Speville B, Frigault MJ, Olszanski AJ, Lam VK, Hyland N, Navenot JM, Fayngerts S, Wolchinsky Z, Broad R, Batrakou D, Pentony MM, Sanderson JP, Gerry A, Marks D, Bai J, Holdich T, Norry E, Fracasso PM. Phase I clinical trial evaluating the safety and efficacy of ADP-A2M10 SPEAR T cells in patients with MAGE-A10+ advanced non-small cell lung cancer. J Immunother Cancer. 2022 Jan;10(1):e003581. doi: 10.1136/jitc-2021-003581. PMID 35086946